CLINICAL TRIAL: NCT07037017
Title: Neurophysiological Effects of Cognitive-Behavioral Therapy in Anorexia Nervosa: A Pre-Post EEG, GSR, and Eye-Tracking Study
Brief Title: CBT Effects on Neural, Physiological, and Attentional Responses in Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Collaborators: Uskudar University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Assistant Professor, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN-CBT-EEG-2025
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorders (Excluding Anorexia Nervosa)
Keywords: Cognitive Behavioral Therapy (CBT); EEG; Eye-Tracking; Galvanic Skin Response (GSR); Body Image
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A two-arm, parallel-group, randomized controlled trial comparing the effects of a 12-week Cognitive-Behavioral Therapy program versus a waitlist control in individuals with restrictive-type anorexia nervosa. Participants undergo neurophysiological (EEG), physiological (GSR), and attentional (eye-tracking) assessments before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Intervention Group (Experimental): Participants diagnosed with restrictive-type anorexia nervosa will receive 12 weekly individual Cognitive-Behavioral Therapy (CBT) sessions. Each session will last approximately 60 minutes and be delivered by a trained therapist. The CBT protocol targets body image distortion, cognitive restructuring of maladaptive beliefs, exposure to food-related stimuli, emotional regulation strategies, and behavioral experiments to reduce avoidance. Pre- and post-treatment neurophysiological (EEG), physiological (GSR), and attentional (eye-tracking) assessments will be conducted.
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Waitlist Control Group (No Intervention): Participants diagnosed with restrictive-type anorexia nervosa will be placed on a waitlist and will not receive any structured psychological intervention during the 12-week study period. They will complete the same neurophysiological (EEG), physiological (GSR), and attentional (eye-tracking) assessments at baseline and at the 12-week follow-up.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Manualized 12-week CBT protocol focused on reducing body image disturbance, distorted beliefs about food and appearance, and avoidance behaviors in individuals with anorexia nervosa. The intervention incorporates psychoeducation, cognitive restructuring, emotional regulation, food exposure, and body image work.
  Arms: CBT Intervention Group

SUMMARY:
This randomized controlled trial investigates the neurophysiological, physiological, and attentional effects of Cognitive-Behavioral Therapy (CBT) in individuals with restrictive-type anorexia nervosa (AN). The study compares two groups: one receiving a 12-week CBT intervention, and one placed on a waitlist (no active treatment during the study period). All participants undergo pre- and post-intervention assessments using electroencephalography (EEG), galvanic skin response (GSR), and eye-tracking while exposed to visual stimuli related to food, body image, and self-appearance. The primary outcomes include neural changes in attention and emotional processing (P300, LPP, frontal alpha asymmetry), physiological arousal (skin conductance), and visual attention biases (fixation duration and gaze distribution). The aim is to determine whether CBT leads to measurable improvements in neurobiological and attentional mechanisms related to body image disturbance and food-related anxiety in AN, contributing to biomarker-informed psychotherapy approaches.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a severe psychiatric disorder characterized by distorted body image, food restriction, and intense fear of weight gain. Despite the effectiveness of Cognitive-Behavioral Therapy (CBT) in targeting maladaptive cognitions and behaviors, its underlying neurophysiological mechanisms remain insufficiently understood. This study aims to evaluate the effects of a 12-week CBT intervention on neural, physiological, and attentional responses in individuals with restrictive-type AN using a randomized controlled trial design.

Sixty female participants (aged 18-35) with restrictive-type AN will be recruited and randomly assigned to one of two groups: a CBT intervention group (n = 30) and a waitlist control group (n = 30). Both groups will undergo baseline and post-intervention assessments using EEG, GSR, and eye-tracking. The CBT intervention will consist of weekly 60-minute sessions for 12 weeks, delivered by trained therapists, and will target body image distortion, cognitive restructuring, exposure to food-related stimuli, emotional regulation, and avoidance behaviors.

During the experimental task, participants will view a series of visual stimuli including (1) self-images (unaltered, altered-thin, altered-overweight), (2) food images (low- vs. high-calorie), and (3) images of other female bodies (thin vs. normal weight). EEG markers of interest include P300 (attentional salience), Late Positive Potential (LPP; sustained emotional reactivity), and frontal alpha asymmetry (indicative of affect regulation and self-referential processing). It is hypothesized that CBT will lead to reductions in P300 and LPP amplitudes and an increase in left-frontal cortical activity, indicating enhanced emotional control and reduced fixation on thin-ideal stimuli.

GSR will be used to assess physiological arousal in response to distressing stimuli. It is expected that post-CBT participants will exhibit lower skin conductance responses (SCRs) to body and food images, indicating improved autonomic regulation. Eye-tracking data will capture fixation durations and gaze patterns. Participants in the CBT group are expected to show less visual attention toward "problematic" body areas (waist, stomach, thighs) and reduced avoidance of high-calorie food images compared to the waitlist group.

Participants will also complete standardized psychometric instruments including the Eating Disorder Examination Questionnaire (EDE-Q), Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), the Yale-Brown Obsessive-Compulsive Scale for Body Dysmorphic Disorder (YBOCS-BDD), and the Cognitive Emotion Regulation Questionnaire (CERQ) at both time points.

This trial will provide critical insights into the neurophysiological and attentional mechanisms of CBT in AN, aiming to identify objective biomarkers of therapeutic change. Results may inform precision-based treatment models and support the development of digitally enhanced or neuromodulation-augmented therapies for eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 35
* Meeting DSM-5 diagnostic criteria for restrictive-type anorexia nervosa
* Body Mass Index (BMI) between 15.0 and 18.5
* Medically stable to participate in psychological and neurophysiological assessments
* Willingness to participate in weekly therapy sessions (for the CBT group) and to complete pre- and post-assessments
* Ability to provide informed consent

Exclusion Criteria:

* Current or past diagnosis of bulimia nervosa, binge-eating disorder, or other eating disorders
* Presence of comorbid severe psychiatric disorders (e.g., psychosis, bipolar disorder, substance use disorder)
* History of neurological illness or traumatic brain injury
* Use of psychotropic medication within the last 6 weeks
* Prior participation in structured Cognitive-Behavioral Therapy for an eating disorder
* Pregnancy
* Visual or neurological impairments that would prevent accurate EEG, GSR, or eye-tracking recordings

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in EEG P300 amplitude in response to body image stimuli | aseline and Week 12
  P300 amplitudes will be extracted from EEG data during visual exposure to body image stimuli. Reduced amplitudes post-CBT are hypothesized to indicate reduced attentional salience and hyperfocus on appearance-related cues. P300 amplitudes will be extracted from EEG data during visual exposure to body image stimuli. Reduced amplitudes post-CBT are hypothesized to indicate reduced attentional salience and hyperfocus on appearance-related cues.
Change in Late Positive Potential (LPP) amplitude to body and food stimuli | Baseline and Week 12
  LPP amplitudes will be measured during viewing of thin, overweight, and food-related images. A reduction post-CBT suggests decreased sustained emotional reactivity to distressing visual input.
Change in frontal alpha asymmetry during self-image viewing | Baseline and Week 12
  Frontal alpha asymmetry (FAA), computed from EEG data, will be used to index emotional regulation. An increase in left-dominant FAA is expected post-CBT, reflecting enhanced emotional control and positive self-perception.
Change in skin conductance response (SCR) to body and food stimuli | Baseline and Week 12
  Skin conductance responses will be measured via GSR during visual exposure to self-body, other-body, and food stimuli. Decreased SCR amplitudes post-CBT will indicate reduced physiological arousal and distress.
Change in fixation duration on weight-related body areas | Baseline and Week 12 Baseline and Week 12
  Eye-tracking will assess gaze fixation duration on areas of interest (waist, thighs, stomach). Post-CBT reductions in fixation on these regions suggest reduced attentional bias toward body dissatisfaction zones.

SECONDARY OUTCOMES:
Change in Eating Disorder Examination Questionnaire (EDE-Q) scores | Baseline and Week 12
  The EDE-Q assesses eating disorder symptoms across four subscales: Restraint, Eating Concern, Weight Concern, and Shape Concern. Each item is rated from 0 (no pathology) to 6 (high pathology). Global score ranges from 0 to 6. Higher scores indicate greater eating pathology. A reduction in post-treatment scores indicates improvement in eating disorder symptoms.
Change in Beck Depression Inventory-II (BDI-II) scores | Baseline and Week 12
  The BDI-II consists of 21 items scored from 0 to 3, yielding a total score between 0 and 63. Higher scores reflect more severe depressive symptoms:
  0-13: minimal 14-19: mild 20-28: moderate 29-63: severe A decrease in BDI-II score post-CBT is expected, reflecting reduced depressive symptoms.
Change in Beck Anxiety Inventory (BAI) scores | Baseline and Week 12
  The BAI includes 21 items rated from 0 to 3, with a total score ranging from 0 to 63. Higher scores indicate more severe anxiety:
  0-7: minimal 8-15: mild 16-25: moderate 26-63: severe Post-CBT reductions in BAI scores suggest improved anxiety regulation.
Change in Yale-Brown Obsessive Compulsive Scale - Body Dysmorphic Disorder Version (YBOCS-BDD) scores | Baseline and Week 12
  The YBOCS-BDD contains 12 items rated from 0 to 4, yielding a total score range of 0 to 48. Higher scores reflect greater severity of body image-related obsessions and compulsions. Scores ≥ 20 are considered moderate to severe. Post-treatment reductions reflect decreased symptom severity.
Change in Cognitive Emotion Regulation Questionnaire (CERQ) scores | Baseline and Week 12
  The CERQ includes 36 items rated from 1 (almost never) to 5 (almost always), across 9 subscales (e.g., catastrophizing, reappraisal, rumination). Subscale scores range from 4 to 20. Higher scores in adaptive subscales and lower scores in maladaptive subscales post-CBT indicate improved emotional coping. The CERQ includes 36 items rated from 1 (almost never) to 5 (almost always), across 9 subscales (e.g., catastrophizing, reappraisal, rumination). Subscale scores range from 4 to 20. Higher scores in adaptive subscales and lower scores in maladaptive subscales post-CBT indicate improved emotional coping.
Change in subjective distress ratings on Visual Analog Scale (VAS) | Immediately after the experimental task at both baseline and Week 12
  The VAS is a self-reported 0-10 scale used to assess momentary emotional distress following exposure to visual stimuli.
  0 = no distress 10 = extreme distress Lower VAS scores after CBT indicate increased emotional tolerance of body and food-related images.

CONTACTS AND LOCATIONS:
Overall Officials: Gökben Hızlı Sayar, Professor, Study Chair — Üsküdar University; Eda Yılmazer, Phd, Study Director — Beykoz University
Locations (1):
- Üsküdar University Neuro Marketing Lab., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for all primary and secondary outcome measures (EEG, GSR, eye-tracking, and psychometric scores) will be shared upon reasonable request. Data will be shared in compliance with institutional ethics and data protection regulations.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD and supporting materials will be available beginning 6 months after publication of the primary results and will remain available for up to 5 years upon request.
Access Criteria: Qualified researchers affiliated with academic institutions may request access to the IPD and supporting materials for ethically approved secondary analyses. Requests must include a brief research proposal and will be reviewed by the study investigators. Data will be shared via secure institutional transfer platforms upon data use agreement. Qualified researchers affiliated with academic institutions may request access to the IPD and supporting materials for ethically approved secondary analyses. Requests must include a brief research proposal and will be reviewed by the study investigators. Data will be shared via secure institutional transfer platforms upon data use agreement.